## **Summary of Statistical Analysis Plan for MYTHIC Study**

[Draft: April 26, 2020]

| Part | Patient Group(s) | Outcome | Statistical Analysis <sup>a</sup> |
|---|---|---|---|
| 1 | Arm 1 (ITT) | SVR12 | - estimated probability of SVR12 and 95% confidence interval (CI) - exact binomial calculations |
| 2 | Arm 1 (ITT) | Virologic failure (VF) | - estimated probability of SVR12 and 95% confidence interval (CI) - exact binomial calculations |
| 3 | Arm 1 (ITT) | Post-treatment virologic relapse | - estimated probability of SVR12 and 95% confidence interval (CI) - exact binomial calculations |
| 4 | All patients | HCV-viremic kidney<br>transplant (KT); i.e.,<br>Arm 1 KT | - cumulative incidence and 95% CI - death and other KT types treated as competing risk - estimate non-parametrically, using Lin (1997) which proceeds through the cause-specific hazards, or Fan (2013) which uses Inverse Probability of Censoring Weighting (IPCW). |
| 5 | All patients | Non-HCV-viremic KT;<br>i.e., Arm 2A-2B KT | - same as for component (4). |
| 6 | All, by Arm | Hospital admissions | - Arm treated as a time-dependent treatment - crude hospitalization rate per 100 patient-years (PY) and 95% CI - use robust variance estimator, to account for correlation among hospital admissions within-patient |
| 7 | All, by Arm | Hospital admissions | - Arm treated as a time-dependent treatment - proportional rates model (Lin et al., 2000) - robust SEs, to account for clustering within-patient |
| 8(a) | All, and SRTR* controls | Kidney transplant | <ul> <li>exclude, from SRTR, all patients who indicated consent to receive an HCV-viremic KT (hereafter: SRTR*)</li> <li>estimate prognostic score using SRTR* patients: KT as event</li> <li>1:5 matching (MYTHIC: SRTR*) based on prognostic score with caliper</li> <li>Cox regression, with MYTHIC as lone covariate, stratified by matched set</li> </ul> |

| 8(b) | All, and SRTR* | Kidney transplant | Same as 9(a), but using exact matching on small set of predictors, with prognostic |
|---|---|---|---|
| | controls | | score used to break ties among potential matches |
| 9 | Arm 1 – ITT | Compliance | Treated as repeated binary (0/1) data, with 1 indicating compliance (i.e., having |
| | | | taken 80-120% of prescribed pills) |
| 10 | Arm 1 – ITT | Death | Time to event; Cox regression |
| 11 | Arm 1 – ITT | Graft failure | Time to event; Cox regression |
| 12 | Arm 1 | Delayed graft | DGF: binary (0/1) response. |
| | | function | Compute OBS/EXP, where OBS=observed number of DGFs for Arm 1 and EXP= |
| | | | expected count based on logistic regression model fitted to HCV-negative UNOS |
| | | | patients from large academic centers |
| 13 | Arm 1 | Acute allograft | AAR: Binary (0/1) response. |
| | | rejection | Compute OBS/EXP, where OBS=observed number of AARs for Arm 1 and EXP= |
| | | | expected cunt based on logistic regression model fitted to HCV-negative UNOS |
| | | | patients from large academic centers |
| 14 | Arm 1 | ALT elevation | Binary (0/1), with '1' corresponding to peak ALT > 5 x ULN, where ULN=upper |
| | | | limit of 'normal'. |
| 15 | All, by arm | Serious Adverse | SAE: recurrent event |
| | | Event | Arm treated as a time-dependent factor |
| | | | Proportional rates model, robust SEs to account for within-patient clustering |
| 16 | Arm 1, 2AB | eGFR | Repeated continuous response |
| | | | Linear mixed model, to account for clustering by patient |
| 17 | Arm 1, 2AB | Proteinuria | Binary response; logistic regression |
| 18 | Arm 1, 2AB | BK virus | Binary response; logistic regression |

## Notes:

a) Each of the above-listed analyses will be accompanied by appropriate summary statistics (e.g., mean, median, IQR, etc).